CLINICAL TRIAL: NCT04849091
Title: Investigating the Clinical Effectiveness of iReadMore; a Digital Therapy for People With Alexia (Acquired Dyslexia)
Brief Title: Clinical Effectiveness of iReadMore for People With Alexia
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University College, London (Other)
Collaborators: Medical Research Council (Other Government)
Responsible Party: Sponsor
Other Study IDs: 7609/001
Record Dates: First submitted 2021-04-07; First posted 2021-04-19 (Actual); Last update posted 2023-05-10 (Actual); Status verified 2023-05

CONDITIONS: Stroke; Brain Injuries; Aphasia; Alexia; Dementia
Keywords: Digital; Therapy; Reading disorder; Alexia; Dyslexia; Rehabilitation
MeSH Terms: conditions — Stroke; Brain Injuries; Aphasia; Dyslexia; Dementia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- iReadMore users: Participants will be iReadMore users who completed a baseline reading test between XX/XX/XXXX and XX/XX/XXXX, and who performed at least 5 hours of reading training and a second (interval) reading test.
  iReadMore users will self-register to participate in the study.
  Interventions: Device: iReadMore

INTERVENTIONS:
Device: iReadMore — Digital Alexia Therapy

SUMMARY:
iReadMore will provide an app-based therapy for people with pure or central alexia.

This study aims to test the clinical effectiveness of iReadMore for improving reading accuracy and speed in real world users of the therapy.

DETAILED DESCRIPTION:
iReadMore is a self-led therapy app for improving single word reading accuracy and speed in individuals with acquired reading impairments. iReadMore has been demonstrated to improve reading speed and accuracy in pure and central alexias (Woodhead et al., 2013, 2018). iReadMore therapy is not expected to improve reading for the remaining alexia subtypes.

iReadMore includes 590 of the most frequently written words from the SUBTLEX lexical database (Brysbaert and New, 2009). High frequency words were chosen to maximise the relevance (ecological utility) of the training to everyday life. The therapy mechanism relies on mass practice of cross-modal, paired associate learning (Holcomb and Anderson, 1993) based on the Triangle Model approach to reading. Untrained words will not be affected, and thus word reading improvements are not expected to generalise beyond trained items.

The therapy utilises gamification and is designed to be accessible in order to drive motivation and engagement for the user group. iReadMore is downloadable via the Google Play store on Android tablet devices. iReadMore is a CE-marked class 1 medical device that was developed by the Neurotherapeutics Group, University College London.

An online roll-out trial will be conducted to evaluate the clinical effectiveness of iReadMore with a study population of real world users. The therapy will be evaluated in a clinical population with a reading impairment of any acquired cause (such as stroke or brain injury). Participants will self-enrol in the study through the app, which has been co-designed to ensure accessibility to this user group.

A within-participant evaluation of trained versus untrained items will investigate the clinical effectiveness of the therapy for improving reading speed and accuracy. The primary outcomes are improvements in single word reading accuracy and speed. Interval testing will be conducted after every 5 hours of therapy. The secondary outcomes are self-reported Activities of Daily Living and a series of qualitative questions.

Further analyses will be conducted on alexia subtypes and the influence of therapy dose and intensity on the therapeutic outcomes.

Ethical approval for the iReadMore roll-out trial was obtained from the UCL Research Ethics Committee (ID: 7609/001).

ELIGIBILITY:
Inclusion Criteria:

* Over 18 years old
* Diagnosed with stroke, dementia, brain injury or brain tumour
* Diagnosed or self-diagnosed with impaired reading ability
* Willing and able to give informed consent for participation in the study

Exclusion Criteria:

* History of developmental reading or speech and language disability

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study involves real world users of the iReadMore therapy who have an acquired reading impairment. Users will self-register into the study via the app. In order to participate, users must have access to WiFi and an Android tablet device.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2021-03-15 (Actual); Primary Completion 2023-12 (Estimated); Study Completion 2024-04 (Estimated)

PRIMARY OUTCOMES:
Word Reading Test - Change in Reading Accuracy and Speed from baseline to 20 hours | At baseline and after every 5 hours of therapy up to a maximum dose of 50 hours. Primary outcome is change from baseline to 20 hours.
  Change in single word reading accuracy and speed will be assessed in a Word Reading Test (WRT) delivered in the app. At interval tests, the WRT will include both trained and untrained words to investigate the treatment-specific effects.

SECONDARY OUTCOMES:
Participant-Reported Outcome Measures - Activities of Daily Living (ADL) | At baseline and after every 10 hours of therapy up to a maximum dose of 50 hours
  Activities of Daily Living - Participants are asked to rate how easy they find completing a series of everyday tasks, including language and non-language related tasks. Responses are reported using a 7-point Likert scale from 0 to 6 denoting 'Very Easy' to 'Very Hard'.
Participant-Reported Outcome Measures - Qualitative Questions | At baseline and after every 10 hours of therapy up to a maximum dose of 50 hours
  Qualitative Questions - participants are also asked three open text questions on their experiences of the therapy and their reading abilities at that point in time.

CONTACTS AND LOCATIONS:
Overall Officials: Alexander P Leff, Professor, Principal Investigator — University College, London
Locations (1):
- Institute of Neurology, University College London, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Woodhead ZVJ, Kerry SJ, Aguilar OM, Ong YH, Hogan JS, Pappa K, Leff AP, Crinion JT. Randomized trial of iReadMore word reading training and brain stimulation in central alexia. Brain. 2018 Jul 1;141(7):2127-2141. doi: 10.1093/brain/awy138. PMID 29912350